CLINICAL TRIAL: NCT06695377
Title: Thromboembolic Complications Post-COVID-19: What is the Risk in Mild-Moderate Cases?
Brief Title: Thromboembolic Complications in Mild Covid-19 Cases
Status: Completed | Type: Observational
Sponsor: Marmara University Pendik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Buğu Usanma Koban, MD, PhD, Marmara University Pendik Training and Research Hospital
Other Study IDs: 02.12.2022.1652
Record Dates: First submitted 2024-11-13; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: COVID 19; Thromboembolic and Bleeding Complications; Thromboembolism, Venous; Post COVID-19
Keywords: COVID 19; thromboembolism; thromboembolic complications; pulmonary embolism; deep venous thrombosis
MeSH Terms: conditions — COVID-19; Venous Thromboembolism; Thromboembolism; Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with a PCR-confirmed COVID-19 diagnosis who were followed up on an outpatient basis

SUMMARY:
The aim of the study is to investigate the frequency of thromboembolic complications and the factors influencing them in COVID-19 cases that did not require hospitalization. For this purpose, patients registered at two different family health centers in Istanbul were retrospectively screened, and their status regarding post-COVID-19 thromboembolic events was recorded. The sociodemographic characteristics, medical history, COVID-19 treatments received, comorbidities, and current medications of all patients were examined and compared with the occurrence of complications.

DETAILED DESCRIPTION:
Studies on COVID-19 complications in the literature have predominantly focused on patients treated in hospitals, particularly in intensive care units. Data on patients with mild to moderate symptoms who were followed up on an outpatient basis in primary care are quite limited. Therefore, our research investigated the incidence of thrombotic events within six months following infection in mild to moderate COVID-19 cases and the factors that might influence these events. Records of 961 individuals registered at two different family health centers in Istanbul were reviewed. Patients were contacted by phone, informed about the study, and data regarding their sociodemographic characteristics, medical histories, COVID-19 infection experiences, and medications used were collected. Comparative analyses (Fisher's exact test) and logistic regression tests were conducted.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Having had a confirmed COVID-19 infection verified by a PCR test
* Being monitored at a family health center without requiring hospitalization during the COVID-19 course
* Having at least 6 months elapsed since the infection
* Availability of the patient's medical records
* Absence of any language barrier or health issue that would prevent communication with the patient

Exclusion Criteria:

* Being under 18 years of age
* Having had less than 6 months since the COVID-19 infection
* Presence of any condition that prevents communication with the patient
* Incomplete or missing medical records of the patient
* History of hospitalization due to COVID-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who were registered at family health centers in two different districts of Istanbul and had a confirmed COVID-19 infection verified by PCR test between January 1, 2022, and June 30, 2022, were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 961 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
The frequency of thromboembolic complications in COVID-19 patients not requiring hospitalization. | january-june 2022
  Patients registered at a family health center were retrospectively reviewed, and those with a history of COVID-19 PCR positivity who had been followed up as outpatients were included. The occurrence of venous or arterial thromboembolism within the first 6 months after infection was recorded from their medical reports, and the frequency was calculated.
The relationship between patients' comorbidities and the occurrence of thromboembolic events post-COVID. | january-june 2022
  The patients' existing chronic conditions from the time of their COVID-19 infection were recorded by reviewing the family medicine system. The presence of chronic diseases was then analyzed in comparison to the occurrence of thrombosis within the first 6 months following COVID-19 infection.
The relationship between patients' medications and the occurrence of thromboembolic events post-COVID. | january-june 2022
  The medications regularly used by patients for their chronic conditions since the time of their COVID-19 infection were noted by reviewing records in the family medicine system. These medications were then analyzed in comparison to the occurrence of thrombosis within the first 6 months following COVID-19 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Buğu Usanma Koban, Principal Investigator — Marmara University Medical Faculty
Locations (1):
- Marmara University Medical School, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The research data may be shared anonymously with researchers if needed.

REFERENCES:
- [Background] Azevedo-Cerqueira A, Torrao Pinheiro P, Oliveira J, Manuel-Marques M, Rocha Neves J. Risk Of Venous Thrombosis In The Primary Care Setting During The Covid-19 Pandemic. Port J Card Thorac Vasc Surg. 2023 Apr 4;30(1):43-47. doi: 10.48729/pjctvs.310. PMID 37029943
- [Background] Katsoularis I, Fonseca-Rodriguez O, Farrington P, Jerndal H, Lundevaller EH, Sund M, Lindmark K, Fors Connolly AM. Risks of deep vein thrombosis, pulmonary embolism, and bleeding after covid-19: nationwide self-controlled cases series and matched cohort study. BMJ. 2022 Apr 6;377:e069590. doi: 10.1136/bmj-2021-069590. PMID 35387772
- [Derived] Usanma Koban B, Celik O, Sur Unal U, Uzuner A. Assessing the Burden of Thromboembolic Complications in Outpatient COVID-19 Cases: A Focused Study on Patients Followed in Primary Care. Can J Infect Dis Med Microbiol. 2025 Jul 24;2025:7242450. doi: 10.1155/cjid/7242450. eCollection 2025. PMID 40747374